CLINICAL TRIAL: NCT00229385
Title: Treatment With Ziprasidone for Schizophrenia Patients With Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Joseph Zohar, Prof. Joseph Zohar, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHEBA-03-3061-JS-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia; Obsessive Compulsive Disorder
MeSH Terms: conditions — Schizophrenia; Obsessive-Compulsive Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Ziprasidone
- 2 (Active Comparator)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — 40-80 mg BID

SUMMARY:
Comparing schizophrenic patients with comorbid OCD and schizophrenic patients without OCD in response to Ziprasidone and in cognitive functioning as compared with OCD patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia and OCD for at least 6 months
* Minimum score of 14 on YBOCS
* Minimum score of 60 on PANSS
* Diagnosis of Schizophrenia without OC symptoms

Exclusion Criteria:

* Patients who are already being treated with ziprasidone
* Diagnosis of schizophreniform disorder
* Organic brain syndrome, mental retardation and pervasive developmental disorder
* Patients having any significantly cardiovascular illness or electrolyte imbalance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
YBOCS | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel